CLINICAL TRIAL: NCT05795361
Title: Post-trial Access Program: Idursulfase-IT (HGT-2310) in Conjunction With Intravenous Elaprase® in Pediatric and Adult Patients With Hunter Syndrome and Cognitive Impairment
Brief Title: Post-trial Access Program of Idursulfase-IT Along With Elaprase in Children With Hunter Syndrome
Status: Available | Type: Expanded Access
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-609-5005
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Hunter Syndrome
MeSH Terms: conditions — Mucopolysaccharidosis II

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Idursulfase-IT — Participants will continue to receive the same dose of idursulfase-IT, once monthly, that was administered during the HGT-HIT-046 [NCT01506141] or SHP609-302 [NCT02412787] study [10mg or 30mg] along with intravenous (IV) infusions of standard-of-care therapy Elaprase via intrathecal drug delivery device (IDDD) or lumbar punctures.
  Other Names: HGT-2310; TAK-609

SUMMARY:
As the HGT-HIT-046 (NCT01506141) and SHP609-302 (NCT02412787) studies will be closed, this post-trial access (PTA) program provides TAK-609 to participants in these studies for whom the benefit:risk ratio of continued treatment with idursulfase-IT remains positive.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will have completed the treatment period of the HGT-HIT-046 (NCT01506141) or SHP609-302 (NCT02412787) study prior to the first dose on this program.
2. Participant and/or a parent(s)/legal guardian is informed of the nature of this compassionate post-trial access program and can provide written informed consent for themselves or the child to participate (with assent from the child when appropriate prior to treatment).

Exclusion Criteria:

1. Participant has a condition that in the opinion of the treating physician may compromise their safety.
2. Participant has a known hypersensitivity to idursulfase-IT or its components.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (22):
- United States (17):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - The Regents of the University of California, Oakland, California
  - The Nemours Foundation, Wilmington, Delaware
  - Jackson Memorial Hospital University of Miami, Miami, Florida
  - Ann and Robert H Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - Washington University, Washington, Missouri
  - Board of Regents of the University of Nebraska, Omaha, Nebraska
  - Joseph M. Sanzari Children's Hospital, Hackensack, New Jersey
  - NYU Langone Medical Center, New York, New York
  - The University of North Carolina, Chapel Hill, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Randall Children's Hospital at Legacy Emanuel, Portland, Oregon
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Childrens Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Division of Medical Genetics, University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital - PIN, Seattle, Washington
- Queensland Childrens Hospital, South Brisbane, Queensland, Australia
- Mexico (2):
  - Instituto Nacional de Pediatria, Coyoacán, Mexico City
  - H.C.U. de Valladolid, Valladolid
- Hospital Universitario Reina Sofia, Córdoba, Spain
- Royal Manchester Children's Hospital - PPDS, Manchester, United Kingdom

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/1a50b2ee12ee4e80?idFilter=%5B%22TAK-609-5005%22%5D